CLINICAL TRIAL: NCT05040503
Title: Monitoring Mitophagy In Myeloid Cells Upon Intensive Care
Acronym: MIMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUENOT 2020-2
Record Dates: First submitted 2021-08-30; First posted 2021-09-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients without sepsis (Active Comparator): patient without sepsis admitted to the Intensive Care Unit or the Anesthesia and Intensive Care Unit of the Dijon University Hospital
  Interventions: Biological: Blood sampling at inclusion; Biological: Blood sampling at 24 hours; Other: Data collection
- Patients with sepsis (Experimental): Patients with sepsis admitted to the Intensive Care Unit or the Anesthesia and Intensive Care Unit of the Dijon University Hospital
  Interventions: Biological: Blood sampling at inclusion; Biological: Blood sampling at 24 hours; Other: Data collection
- Patients with septic shock (Experimental): Patients with septic shock admitted to the Intensive Care Unit or the Anesthesia and Intensive Care Unit of the Dijon University Hospital
  Interventions: Biological: Blood sampling at inclusion; Biological: Blood sampling at 24 hours; Other: Data collection
- Healthy volunteers (Active Comparator)
  Interventions: Biological: Blood sampling at inclusion; Other: Data collection

INTERVENTIONS:
Biological: Blood sampling at inclusion — Sampling of 2 tubes of 3 ml:
  * patient: H0: 0-6h post-admission
  * healthy volunteer: at inclusion
Biological: Blood sampling at 24 hours — Collection of 2 tubes of 3 ml (H24: 24-30h post-admission)
  Arms: Patients with sepsis; Patients with septic shock; Patients without sepsis
Other: Data collection — clinical and biological medical data for patients and general health data for healthy volunteers

SUMMARY:
Severe infections (sepsis) are a frequent cause of admission to the intensive care unit. Sepsis represent a significant risk for the health of patients in the short and medium term. Sepsis are notably linked to a change in the function of immune cells. In some patients, a state of pseudo-dormancy of monocyte and macrophage immune cells, called myeloid cell immunosuppression, is observed. This situation, which leads to a worsening of the infection, must be avoided because it represents a danger for the patient, even during antibiotic therapy. At present, these events are still very poorly understood. Research is needed to understand how the immunosuppression of myeloid cells occurs in order to adapt existing treatments or to find new ones.

Laboratory work on animal models of sepsis has shown that this state of myeloid cell immunosuppression is closely linked to a modification of energy production by myeloid cells (monocytes and macrophages). The function of the mitochondria ("energy factory" of the cells) in these cells is impaired. Thus, restoring mitochondrial function in myeloid cells could be a therapeutic solution against the immunosuppression of myeloid cells during severe sepsis.

The aim of this study is to verify whether alterations in mitochondrial function in myeloid cells occur in both patients with and without bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to all 4 groups:

* Patient (and/or trusted person/health care proxy or relative) or volunteer who provided oral consent after receiving information about the study, or patient included in emergency situation
* Age ≥ 18 years

Common criteria for patients

- Admission to the Intensive Care Unit or the Anesthesia and Intensive Care Unit of the Dijon University Hospital

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person subject to a measure of legal protection (curatorship, guardianship)
* Person subject to limited judicial protection
* Pregnancy or breastfeeding
* Known primary or secondary immune deficiency (radiotherapy, chemotherapy, immunosuppressive treatment or systemic corticosteroid therapy in the 3 months preceding inclusion (> 0.15 mg/kg/d of prednisone equivalent for more than 2 weeks or "bolus" greater than 2mg/kg/d of prednisone equivalent), HIV infection, primary cellular immune deficiency)
* Patients hospitalized within 3 months prior to inclusion for sepsis.
* Patients receiving therapy known to modulate mitochondrial function, mitochondrial biogenesis or mitophagy (chloroquine, hydroxychloroquine, rapamycin, carbamazepine, resveratrol, sildenafil)
* Patients with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Level of mitophagy | at admission and at 24 hours post-admission

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No